CLINICAL TRIAL: NCT01317420
Title: A Phase I Dose Escalation Trial of BI 836845 Administered Intravenously Once Every Three Weeks in Patients With Advanced Solid Tumours During Escalation and Weekly in Selected Tumour Types During Expansion, With Repeated Administrations in Patients Showing Clinical Benefit
Brief Title: Trial to Determine MTD of BI 836845 Administered Intravenously Once Every Three Weeks in Patients With Advanced Solid Tumours and Later a Weekly Dosing Schedule in Selected Tumour Types
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1280.2; 2010-021714-29 (EudraCT Number)
Record Dates: First submitted 2011-03-15; First posted 2011-03-17 (Estimated); Results first posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — xentuzumab

ARMS (13):
- BI 836845 10 mg (Experimental): Patients received 10 milligram (mg) of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
  Interventions: Drug: BI 836845
- BI 836845 20 mg (Experimental): Patients received 20 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
  Interventions: Drug: BI 836845
- BI 836845 40 mg (Experimental): Patients received 40 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
  Interventions: Drug: BI 836845
- BI 836845 80 mg (Experimental): Patients received 80 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
  Interventions: Drug: BI 836845
- BI 836845 160 mg (Experimental): Patients received 160 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
  Interventions: Drug: BI 836845
- BI 836845 320 mg (Experimental): Patients received 320 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
  Interventions: Drug: BI 836845
- BI 836845 640 mg (Experimental): Patients received 640 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
  Interventions: Drug: BI 836845
- BI 836845 1280 mg (Experimental): Patients received 1280 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
  Interventions: Drug: BI 836845
- BI 836845 1800 mg (Experimental): Patients received 1800 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
  Interventions: Drug: BI 836845
- BI 836845 2400 mg (Experimental): Patients received 2400 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
  Interventions: Drug: BI 836845
- BI 836845 3600 mg (Experimental): Patients received 3600 mg of BI 836845 (concentrate for solution for infusion) given intravenously for 1 hour on Day 1 of each 3-weekly course of treatment until disease progression or undue toxicities in the dose escalation part of the study
  Interventions: Drug: BI 836845
- Ewings sarcoma (Experimental): Patients with Ewing's family of tumours (EFT) or primitive neuroectodermal tumour (PNET) receiving relevant biological dose (RBD) of BI 836845 1000 mg, administered in each course of 21 days by a 1-hour infusion at the start of each week in expansion part of the study.
  Interventions: Drug: BI 836845
- Biopsiable tumours (Experimental): Patients with all solid tumour types who had tumours suitable for biopsy receiving relevant biological dose (RBD) of BI 836845 1000 mg, administered in each course of 21 days by a 1-hour infusion at the start of each week in expansion part of the study.
  Interventions: Drug: BI 836845

INTERVENTIONS:
Drug: BI 836845 — Intravenous infusion
  Other Names: Xentuzumab

SUMMARY:
This study is a phase I, open-label, dose escalation trial to determine the maximum tolerated dose (MTD) of a new drug BI 836845 which blocks the insulin growth factor (IGF) pathway believed to be involved in cancer growth. BI 836845 will be administered for the very first time into cancer patients.

The study will also look at the overall safety of the drug, and examine the drug levels in the body at specific timepoints during the trial (pharmacokinetic profile); the effect the drug may have on tumours will also be examined (pharmacodynamics).

ELIGIBILITY:
Inclusion criteria:

1. Male or female patients with cytologically or histologically confirmed solid tumours that are refractory to standard therapy or that have no standard therapy.
2. Patients should have evaluable disease, or at least one measurable lesion according to Response Evaluation Criteria In Solid Tumours (RECIST) criteria version 1.1
3. Age, equal, or more than, 18 years old.
4. Life expectancy of at least 3 months.
5. Written informed consent that is consistent with ICH-GCP guidelines.
6. Eastern Cooperative Oncology Group (ECOG) performance score 0, 1 or 2.
7. Patients must have recovered from any previous surgery and no major surgery within the last 28 days prior to start of trial medication.
8. Cardiac left ventricular function with resting ejection fraction >50% as determined by Echocardiography (ECHO) or Multiple Gated Acquisition scan (MUGA).
9. Absolute neutrophil count equal, or more than, 1,500/µl.
10. Platelets equal, or more than, 100,000/µl.
11. Total bilirubin equal, or less than 1.5 x institution upper limit of normal.
12. Aspartate Amino Transferase (AST) (Serum glutamic oxaloacetic transaminase (SGOT)) / Alanine Amino Transferase (ALT) (Serum glutamic pyruvic transaminase (SGPT )) equal, or less than, 2.5 x upper limit of normal (in case of known liver metastases AST and/or ALT, equal, or less than, 5 x upper limit of normal).
13. Creatinine equal, or less than, 1.5 x institution upper limit of normal.
14. Haemoglobin equal, or more than, 9g/dL.
15. Haemoglobin A1c less than 8% and fasting glucose, equal, or less than, 8.9 mmol/L (= 160 mg/dL).
16. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) for the duration of trial participation. Female patients with reproductive potential must have a negative serum pregnancy test within 7 days of trial enrolment.
17. Patients entering part II of the study should have cytologically or histologically confirmed disease from the Ewing's family of tumours/PNET (cohort 1), or solid tumours suitable for biopsy (cohort 2), that are refractory to standard therapy or that have no standard therapy.
18. Patients eligible to undergo biopsy should have normal coagulation parameters (INR and PTT within normal ranges) and platelet count (equal, or more than, 100,000/µl) prior to biopsy tissue collection.

Exclusion criteria:

1. Active infectious disease.
2. Serious illness or concomitant non-oncological disease considered by the investigator to be incompatible with the protocol.
3. History of thrombosis within 1 year of study or if concurrent anticoagulation required.
4. Patients not recovered from any therapy-related toxicities from previous chemo-, hormone-, immuno-, molecular targeted, or radiotherapies to at least Common Terminology Criteria for Adverse Events (CTCAE) equal, or less than, Grade 1. Prior chemotherapy is allowed if completed at least 4 weeks prior to first trial treatment (6 weeks for mitomycin C or nitrosoureas) and the patient has recovered from the acute toxicities of that therapy.
5. Patients with untreated or symptomatic brain metastases. Patients with treated, asymptomatic brain metastases are eligible if there has been no change in brain disease status for at least 4 weeks before starting trial medication, no history of cerebral oedema or bleeding in the past 4 weeks before starting trial medication and must be on a stable or reducing dose of dexamethasone. Anti-epileptic therapy will be allowed if the patient is stable on antiepileptic treatment for 4 weeks, or more, without adjustments before starting trial medication.
6. Patients who have been treated with any of the following within 4 weeks of starting trial medication: chemotherapy, immunotherapy, radiotherapy, biological therapies (including trastuzumab), molecular targeted, hormone therapy for breast cancer within 2 weeks of starting trial medication (excluding Luteinizing-hormone-releasing hormone (LHRH) agonists in prostate cancer, or bisphosphonates), or treatment with other investigational drugs.
7. Use of any investigational drug within 4 weeks before start of therapy or concomitantly with this trial.
8. Patients unable to comply with the protocol.
9. Active alcohol abuse or active drug abuse (at the discretion of the investigator).
10. Patients with unstable arrhythmias or unstable angina or severe obstructive pulmonary disease within the last year.
11. For patients entering part II of the study, prior use of any insulin growth factor (IGF) inhibitor.
12. Patients with a history of diabetes mellitus.
13. Pregnancy or breast feeding.
14. Patients that are to undergo biopsy should not have a history of a hereditary bleeding disorder as judged by the investigator.
15. Patients that are to undergo biopsy should pause acetylsalicylic acid treatment for at least 7 days prior to biopsy tissue collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2011-04-13 (Actual); Primary Completion 2016-02-15 (Actual); Study Completion 2016-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- United Kingdom (2):
  - St James's University Hospital, Leeds
  - The Royal Marsden Hospital, Sutton, Sutton

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] de Bono J, Lin CC, Chen LT, Corral J, Michalarea V, Rihawi K, Ong M, Lee JH, Hsu CH, Yang JC, Shiah HS, Yen CJ, Anthoney A, Jove M, Buschke S, Fuertig R, Schmid U, Goeldner RG, Strelkowa N, Huang DC, Bogenrieder T, Twelves C, Cheng AL. Two first-in-human studies of xentuzumab, a humanised insulin-like growth factor (IGF)-neutralising antibody, in patients with advanced solid tumours. Br J Cancer. 2020 Apr;122(9):1324-1332. doi: 10.1038/s41416-020-0774-1. Epub 2020 Mar 12. PMID 32161368
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open label, uncontrolled, dose escalation, 3+3 design, and multicenter study in two parts. Part 1: dose escalation in patients with advanced solid tumours to determine the MTD or RBD. Part 2: expansion part at the RBD in patients with selected tumour types more likely to benefit from BI 836845 (Cohort 1- Ewing's family of tumours or PNET; Cohort 2 - biopsiable solid tumours) in order to investigate safety and PK/pharmacodynamics.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | BI 836845 10 mg | BI 836845 20 mg | BI 836845 40 mg | BI 836845 80 mg | BI 836845 160 mg | BI 836845 320 mg | BI 836845 640 mg | BI 836845 1280 mg | BI 836845 1800 mg | BI 836845 2400 mg | BI 836845 3600 mg | Ewings Sarcoma | Biopsiable Tumours
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 11 | 20
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 11 | 20
Not completed — Progressive disease according to RECIST | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 11 | 16
Not completed — Other adverse event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Non-compliant with protocol | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Refused to cont. taking trial medication | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Reason other than those specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set: All enrolled patients who gave informed consent and who were documented to have taken at least one dose of investigational treatment. The treated set was used for all planned analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 836845 10 mg | BI 836845 20 mg | BI 836845 40 mg | BI 836845 80 mg | BI 836845 160 mg | BI 836845 320 mg | BI 836845 640 mg | BI 836845 1280 mg | BI 836845 1800 mg | BI 836845 2400 mg | BI 836845 3600 mg | Ewings Sarcoma | Biopsiable Tumours | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 11 | 20 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (16.3) | 55.7 (20.6) | 56.0 (11.1) | 39.0 (17.4) | 63.0 (14.4) | 43.0 (17.3) | 51.0 (20.0) | 46.3 (14.6) | 64.0 (1.0) | 66.3 (12.5) | 63.7 (8.1) | 29.7 (9.2) | 60.3 (10.7) | 52.5 (16.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 2 | 1 | 2 | 1 | 1 | 2 | 0 | 1 | 2 | 3 | 8 | 24
  Male | 3 | 2 | 1 | 2 | 1 | 2 | 2 | 1 | 3 | 2 | 1 | 8 | 12 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 11 | 20 | 64
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 2 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 11 | 20 | 62
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) or Relevant Biological Dose (RBD) of BI 836845 During the First Treatment Course of the Dose Escalation Phase
Description: To determine the MTD or relevant biological dose (RBD) of BI 836845 during the first treatment course of the dose escalation phase. The MTD was defined as the highest dose level of BI 836845 below the maximum dose administered at which no more than 1 out of 6 patients experienced a drug-related DLT during the first course of treatment. Starting dose of 10 mg BI 836845, administered once every 3 weeks. Dose levels evaluated were: 10 mg, 20 mg, 40 mg, 80 mg, 160 mg, 320 mg, 640 mg, 1280 mg, 1800 mg, 2400 mg, and 3600 mg. In the absence of the MTD, the RBD, where a plateau in total Insulin-like growth factor 1 (IGF-1) level and total neutralisation of IGF activity is predicted, is reported.
Time Frame: During the first course of treatment, up to 21 days
Population: Treated set (TS) restricted to part 1 - dose escalation phase: All enrolled patients who gave informed consent and who were documented to have taken at least one dose of investigational treatment in the dose escalation phase.
Measure: Number; unit: mg
Groups:
- BI 836845: BI 836845 administered intravenously once every three weeks in patients with advanced solid tumours during dose escalation part of the study
Arm/Group | BI 836845
Number analyzed (Participants) | 33
mg | 1000

2. Primary Outcome: Percentage of Patients With Dose Limiting Toxicities (DLTs) During the First Treatment Course of the Dose Escalation Phase
Description: DLTs defined as drug related: CTCAE Grade 4 neutropenia lasting ≥7 days; febrile neutropenia and/or documented infection with Absolute Neutrophil Count <1.0x109/L; Grade 4 thrombocytopaenia or Grade 3 associated with bleeding needing platelet transfusion; Grade ≥3 increased hepatic enzymes; Grade 3 or 4 non-haematologic toxicity with exceptions; Grade ≥2 infusion reaction despite adequate pre-medication; Grade ≥2 nausea and/or vomiting persisting for ≥7 days despite antiemetic treatment; Grade ≥3 skin toxicity despite adequate supportive care measures for up to 2 weeks if it does not reach an improvement to grade ≤2; Grade ≥3 hyperglycaemia resistant to treatment with anti-diabetic agents; any electrolyte grade 3 AE refractory to optimal correction therapy; no recovery from a non-DLT grade >2 toxicity to grade 1 within 14 days of administered dose; sustained fatigue/asthenia grade 3 for >96 h associated with deterioration of Performance score (Eastern Cooperative Oncology Group).
Time Frame: During the first course of treatment, up to 21 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | BI 836845 10 mg | BI 836845 20 mg | BI 836845 40 mg | BI 836845 80 mg | BI 836845 160 mg | BI 836845 320 mg | BI 836845 640 mg | BI 836845 1280 mg | BI 836845 1800 mg | BI 836845 2400 mg | BI 836845 3600 mg
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3
percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Best Overall Response Based on Response Evaluation Criteria In Solid Tumours (RECIST) Criteria Version 1.1
Description: Best overall response (complete response [CR], partial response [PR], stable disease [SD], progressive disease [PD]) based on RECIST criteria version 1.1:
  CR for target lesions: Disappearance of all target lesions. CR for non-target lesions: Disappearance of all non-target lesions and normalization of tumour marker level. All lymph nodes must be non-pathological in size (<10 millimeters [mm] short axis).
  PR: At least a 30% decrease in the sum of diameters (SoD) of target lesions taking as reference the baseline sum diameters.
  SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as references the smallest SoD while on study.
  PD: At least a 20% increase in the sum of the diameters (SoD) of target lesions taking as reference the smallest SoD recorded since the treatment started, together with an absolute increase in the SoD of at least 5 mm; Appearance of 1 or more new lesions; Unequivocal progression of existing non-target lesions.
Time Frame: First treatment administration, up to 246 days.
Population: TS
Measure: Number; unit: Percentage of participants
Arm/Group | BI 836845 10 mg | BI 836845 20 mg | BI 836845 40 mg | BI 836845 80 mg | BI 836845 160 mg | BI 836845 320 mg | BI 836845 640 mg | BI 836845 1280 mg | BI 836845 1800 mg | BI 836845 2400 mg | BI 836845 3600 mg | Ewings Sarcoma | Biopsiable Tumours
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 11 | 20
Percentage of participants
  CR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SD | 33 | 33 | 0 | 0 | 0 | 33 | 33 | 33 | 67 | 67 | 33 | 36 | 45
  PD | 67 | 33 | 100 | 100 | 100 | 67 | 67 | 33 | 33 | 33 | 67 | 55 | 25
  Not evaluable | 0 | 33 | 0 | 0 | 0 | 0 | 0 | 33 | 0 | 0 | 0 | 9 | 30

4. Secondary Outcome: Objective Tumour Response
Description: Objective response was defined as best overall response of CR or PR (with no confirmation required).
Time Frame: First treatment administration, up to 246 days.
Population: TS
Measure: Number; unit: Percentage of participants
Arm/Group | BI 836845 10 mg | BI 836845 20 mg | BI 836845 40 mg | BI 836845 80 mg | BI 836845 160 mg | BI 836845 320 mg | BI 836845 640 mg | BI 836845 1280 mg | BI 836845 1800 mg | BI 836845 2400 mg | BI 836845 3600 mg | Ewings Sarcoma | Biopsiable Tumours
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 11 | 20
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Duration of Objective Response
Description: Duration of objective response (days), defined as time from first objective response to the time to progression or death and was only calculated for patients with an objective response (with no confirmation required).
Time Frame: First treatment administration, up to 246 days.
Population: TS. Only participants with objective response were included in the endpoint.
Arm/Group | BI 836845 10 mg | BI 836845 20 mg | BI 836845 40 mg | BI 836845 80 mg | BI 836845 160 mg | BI 836845 320 mg | BI 836845 640 mg | BI 836845 1280 mg | BI 836845 1800 mg | BI 836845 2400 mg | BI 836845 3600 mg | Ewings Sarcoma | Biopsiable Tumours
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Disease Control
Description: Disease control was defined as best overall response of CR, PR (confirmation was not required for CR or PR) or confirmed SD (i.e. lasting for at least 24 weeks).
Time Frame: First treatment administration, up to 246 days.
Population: TS
Measure: Number; unit: Percentage of participants
Arm/Group | BI 836845 10 mg | BI 836845 20 mg | BI 836845 40 mg | BI 836845 80 mg | BI 836845 160 mg | BI 836845 320 mg | BI 836845 640 mg | BI 836845 1280 mg | BI 836845 1800 mg | BI 836845 2400 mg | BI 836845 3600 mg | Ewings Sarcoma | Biopsiable Tumours
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 11 | 20
Percentage of participants | 0 | 0 | 0 | 0 | 0 | 33 | 0 | 0 | 0 | 33 | 0 | 0 | 0

7. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was evaluated in expansion phase of the study. PFS was defined as the time from first treatment administration until tumour progression according to RECIST 1.1 or death from any cause, whichever occurred earlier.
Time Frame: First treatment administration until tumour progression or death, up to 162 days.
Population: Treated set (TS) restricted to part 2 - dose expansion phase: All enrolled patients who gave informed consent and who were documented to have taken at least one dose of investigational treatment in the dose expansion phase.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ewings Sarcoma | Biopsiable Tumours
Number analyzed (Participants) | 10 | 14
days | 37.0 [30.0 to 86.0] | 79.0 [36.0 to 85.0]

8. Secondary Outcome: Maximum Measured Concentration of the Analyte (BI 836845) in Plasma (Cmax)
Description: Maximum measured concentration of the analyte in plasma (Cmax) in the first cycle of treatment (dose escalation phase, part 1) and in the first 3 cycles of treatment (dose expansion phase, part 2).
Time Frame: Part 1: 5 minutes before and 0.5, 1, 2, 4, 7, 24, 72, 168 and 336 h after infusion for Course 1. Part 2: 5 minutes before and 1, 2, 4, 7, 24, 168, 169, 336, 337 h after infusion for Course 1, 2 and 3.
Population: Pharmacokinetic (PK) set: All patients in the treated set who were documented to have received at least one dose of BI 836845 and who had at least one valid PK parameter concentration available. PK data are reported based on the dosage administered to patients.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (µg/mL)
Groups:
- Course 1: Patients are administered BI 836845 weekly in course of 21 days by a 1-hour infusion at the start of each week during course 1 (in expansion part of study)
- Course 2: Patients are administered BI 836845 weekly in course of 21 days by a 1-hour infusion at the start of each week during course 2 (in expansion part of study)
- Course 3: Patients are administered BI 836845 weekly in course of 21 days by a 1-hour infusion at the start of each week during course 3 (in expansion part of study)
Arm/Group | BI 836845 10 mg | BI 836845 20 mg | BI 836845 40 mg | BI 836845 80 mg | BI 836845 160 mg | BI 836845 320 mg | BI 836845 640 mg | BI 836845 1280 mg | BI 836845 1800 mg | BI 836845 2400 mg | BI 836845 3600 mg | Course 1 | Course 2 | Course 3
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 30 | 20 | 10
microgram/milliliter (µg/mL) | 2.45 (10.6) | 5.24 (46.1) | 10.7 (65.8) | 17.7 (17.9) | 66.2 (113) | 196 (163) | 146 (47.8) | 421 (30.8) | 727 (101) | 554 (11.5) | 1080 (10.3) | 295 (19.9) | 399 (26.7) | 419 (26.5)

9. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC)
Description: Area under the plasma concentration-time curve (AUC) of the analyte (BI 836845); AUC(0-504) in part 1 using 3- weekly dosing and AUC(0-168) in part 2 using weekly dosing.
Time Frame: as for outcome 8
Population: PK set. Only participants with available PK data are included in the analysis. PK data are reported based on the dosage administered to patients.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/milliliter (µg*h/mL)
Arm/Group | BI 836845 10 mg | BI 836845 20 mg | BI 836845 40 mg | BI 836845 80 mg | BI 836845 160 mg | BI 836845 320 mg | BI 836845 640 mg | BI 836845 1280 mg | BI 836845 1800 mg | BI 836845 2400 mg | BI 836845 3600 mg | Course 1 | Course 2 | Course 3
Number analyzed (Participants) | 2 | 3 | 3 | 3 | 3 | 3 | 3 | 2 | 3 | 3 | 3 | 27 | 18 | 8
microgram*hour/milliliter (µg*h/mL) | 363 (1.79) | 724 (26.8) | 993 (30.9) | 1910 (50.5) | 5270 (21.6) | 12100 (27.6) | 17300 (61.7) | 34600 (68.2) | 42100 (6.55) | 78500 (6.32) | 87800 (24.9) | 24100 (22.1) | 37300 (33.3) | 36900 (41.6)

10. Secondary Outcome: Time to Maximum Measured Concentration of the Analyte (BI 836845) in Plasma (Tmax)
Description: Time to maximum measured concentration of the analyte in plasma (tmax) in the first cycle of treatment (dose escalation phase, part 1) and in the first 3 cycles of treatment (dose expansion phase, part 2).
Time Frame: as for outcome 8
Population: PK set. PK data are reported based on the dosage administered to patients.
Measure: Median (Full Range); unit: hours
Arm/Group | BI 836845 10 mg | BI 836845 20 mg | BI 836845 40 mg | BI 836845 80 mg | BI 836845 160 mg | BI 836845 320 mg | BI 836845 640 mg | BI 836845 1280 mg | BI 836845 1800 mg | BI 836845 2400 mg | BI 836845 3600 mg | Course 1 | Course 2 | Course 3
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 30 | 20 | 10
hours | 2.2 (10.6) [0.9 to 4.0] | 2.0 (46.1) [1.3 to 2.1] | 1.0 (65.8) [1.0 to 2.1] | 2.1 (17.9) [1.0 to 3.9] | 1.0 (113) [0.5 to 2.0] | 2.0 (163) [1.0 to 2.0] | 2.0 (47.8) [2.0 to 4.0] | 2.3 (30.8) [2.0 to 4.0] | 2.0 (101) [0.9 to 2.0] | 4.0 (11.5) [2.3 to 6.7] | 1.8 (10.3) [1.8 to 3.0] | 2.5 (19.9) [0.9 to 7.0] | 3.0 (26.7) [0.9 to 7.0] | 1.0 (26.5) [0.9 to 4.9]

11. Secondary Outcome: Incidence and Intensity of Adverse Events (AEs) According to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE)
Description: Percentage of patients with adverse events (AEs) according to the grading as per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03, 14 June 2010 are presented.
  When no CTCAE grading was available for a specific event, the intensity of the AE was judged based on the following:
  * Grade 1 - Mild AE; awareness of sign(s) or symptom(s) which were easily tolerated.
  * Grade 2 - Moderate AE; enough discomfort to cause interference with usual activity.
  * Grade 3 - Severe AE; incapacitating or causing inability to work or to perform usual activities.
  * Grade 4 - Life-threatening or disabling AE.
  * Grade 5 - Death related to AE.
Time Frame: From first drug administration, until 21 days after last drug administration, up to 253 days.
Population: TS
Measure: Number; unit: Percentage of participants
Arm/Group | BI 836845 10 mg | BI 836845 20 mg | BI 836845 40 mg | BI 836845 80 mg | BI 836845 160 mg | BI 836845 320 mg | BI 836845 640 mg | BI 836845 1280 mg | BI 836845 1800 mg | BI 836845 2400 mg | BI 836845 3600 mg | Ewings Sarcoma | Biopsiable Tumours
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 11 | 20
Percentage of participants
  Grade 1 | 66.7 | 0.0 | 33.3 | 33.3 | 33.3 | 0.0 | 0.0 | 33.3 | 33.3 | 33.3 | 0.0 | 18.2 | 25.0
  Grade 2 | 0.0 | 33.3 | 33.3 | 0.0 | 33.3 | 0.0 | 66.7 | 33.3 | 0.0 | 33.3 | 66.7 | 45.5 | 45.0
  Grade 3 | 0.0 | 66.7 | 33.3 | 66.7 | 33.3 | 100.0 | 0.0 | 33.3 | 66.7 | 33.3 | 33.3 | 27.3 | 30.0
  Grade 4 | 33.3 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 33.3 | 0.0 | 0.0 | 0.0 | 0.0 | 9.1 | 0.0
  Grade 5 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: From first drug administration, until 21 days after last drug administration, up to 253 days.
Description: Treated set: All enrolled patients who gave informed consent and who were documented to have taken at least one dose of investigational treatment. The treated set was used for all planned analyses.
Groups:
- Ewings Sarcoma: Patients with Ewing's family of tumours (EFT) or primitive neuroectodermal tumour (PNET) receiving relevant biological dose (RBD) of BI 836845 1000 mg, administered in each course of 21 days by a 1- hour infusion at the start of each week in expansion part of the study.
Arm/Group | BI 836845 10 mg | BI 836845 20 mg | BI 836845 40 mg | BI 836845 80 mg | BI 836845 160 mg | BI 836845 320 mg | BI 836845 640 mg | BI 836845 1280 mg | BI 836845 1800 mg | BI 836845 2400 mg | BI 836845 3600 mg | Ewings Sarcoma | Biopsiable Tumours
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 0/3 | 1/3 | 0/3 | 3/3 | 1/3 | 1/3 | 1/3 | 0/3 | 0/3 | 5/11 | 10/20
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 3/3 | 2/3 | 2/3 | 3/3 | 3/3 | 11/11 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI 836845 10 mg (N=3) | BI 836845 20 mg (N=3) | BI 836845 40 mg (N=3) | BI 836845 80 mg (N=3) | BI 836845 160 mg (N=3) | BI 836845 320 mg (N=3) | BI 836845 640 mg (N=3) | BI 836845 1280 mg (N=3) | BI 836845 1800 mg (N=3) | BI 836845 2400 mg (N=3) | BI 836845 3600 mg (N=3) | Ewings Sarcoma (N=11) | Biopsiable Tumours (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspergillus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device dislocation (Product Issues) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 836845 10 mg (N=3) | BI 836845 20 mg (N=3) | BI 836845 40 mg (N=3) | BI 836845 80 mg (N=3) | BI 836845 160 mg (N=3) | BI 836845 320 mg (N=3) | BI 836845 640 mg (N=3) | BI 836845 1280 mg (N=3) | BI 836845 1800 mg (N=3) | BI 836845 2400 mg (N=3) | BI 836845 3600 mg (N=3) | Ewings Sarcoma (N=11) | Biopsiable Tumours (N=20)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 5
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Eustachian tube obstruction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 3
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 3 | 2 | 1 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Gingival erythema (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 2 | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 3 | 8
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 3 | 4
Catheter site erythema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Crepitations (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 1 | 2 | 0 | 0 | 1 | 2 | 1 | 0 | 2 | 1 | 14
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infusion site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal dryness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Suprapubic pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Candiduria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 5
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 3 | 2 | 1 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 2 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nipple pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 3 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.